CLINICAL TRIAL: NCT06456138
Title: Trametinib Plus Anlotinib Combined With Tislelizumab in KRAS-mutant Advanced Non-small Cell Lung Cancer Patients: a Multi-center, Open-label, Phase 1/2 Study
Brief Title: Trametinib Plus Anlotinib Combined With Tislelizumab in KRAS-mutant NSCLC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: BeiGene (Industry); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Baohui Han, Professor, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATT-RAS-001
Record Dates: First submitted 2024-06-05; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: KRAS Mutation-Related Tumors; Advanced Lung Cancer; Refractory Tumor
Keywords: KRAS-mutant NSCLC; Trametinib; Anlotinib; Tislelizumab
MeSH Terms: conditions — Neoplasms | interventions — trametinib; anlotinib; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trametinib + Anlotinib + Tislelizumab (Experimental): In Phase I, there are four treatment arms: anlotinib (6 mg) plus trametinib (1 mg) plus tislelizumab (200 mg, Q3W),
  anlotinib (6 mg) plus trametinib (2 mg) plus tislelizumab (200 mg, Q3W),
  anlotinib (8 mg) plus trametinib (1 mg) plus tislelizumab (200 mg, Q3W),
  and anlotinib (8 mg) plus trametinib (2 mg) plus tislelizumab (200 mg, Q3W).
  In Phase II, there is one treatment arm including trametinib (RP2D) plus anlotinib (RP2D) plus tislelizumab (200 mg, Q3W).
  Interventions: Drug: Trametinib; Drug: Anlotinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Trametinib — Trametinib will be administrated orally every day.
Drug: Anlotinib — Anlotinib will be administrated orally from day 1 to day 14 per 21-day cycle.
Drug: Tislelizumab — Tislelizumab will be administered at full dose (200mg, Q3W) on the patient who received the efficacy evaluation of stable disease (SD) or partial response (PR) or complete response (CR) after 2 cycles' treatment of trametinib plus anlotinib.

SUMMARY:
Lung cancer is the most common cause of cancer-related death worldwide. Approximately 85% to 90% of lung cancer cases are non-small cell lung cancer (NSCLC), of which KRAS is one of the most common driver genes, occurring in 25-30% of lung adenocarcinomas and 3-5% of squamous cell carcinomas. KRAS-mutant NSCLC had been considered undruggable in past decades. This research sought to address a significant challenge in treating NSCLC with KRAS mutations, which are notoriously difficult to target effectively. Here, we proposal that the combined use of anlotinib and trametinib combined with tislelizumab may form an effective strategy for the treatment of KRAS-mutant NSCLC patients.

DETAILED DESCRIPTION:
This is a phase 1/2, open-label, multi-center study aimed at exploring the potential therapeutic efficacy of tislelizumab (intravenous), trametinib (oral) and anlotinib (oral) in KRAS-mutant advanced non-small cell lung cancer patients. The primary objectives were safety, recommended phase 2 dose (RP2D) in Phase I and PFS in Phase II. The secondary aim of the study is to evaluate the progression-free survival (PFS), overall survival (OS), adverse events (AEs), and duration of response (DOR) of the combined strategy in these patients. If the RP2D is reached in Phase I, Phase II will be started; if RP2D is not reached in Phase I, Phase II will not be started. The number of subjects is determined according to the actual situation of dose climbing. All patients will be of histo- and/or cytopathology confirmed. Determination of the KRAS mutation type will be performed in the pathological department of Shanghai Chest Hospital, Shanghai Jiao Tong University School of Medicine. Both ARMS method or targeted sequencing are acceptable. It is not acceptable for subjects with the presence of other driver gene mutation. All eligible subjects must have adequate renal, hepatic, and hematologic function, as defined in "inclusion criteria".

ELIGIBILITY:
Inclusion Criteria:

1. According to the 8th edition of the AJCC/UICC TNM staging system for NSCLC, patients with locally advanced (stage III B/III C), metastatic or recurrent (stage IV) NSCLC confirmed by histology or cytology who are unable to undergo surgery and radical concomitant radiochemotherapy and are confirmed to have at least one measurable lesion according to RECIST 1.1.
2. KRAS mutation positive detected by ARMS or NGS;
3. Have been treated with 1st line of standard therapy and experienced disease progression;
4. Patients who were assessed as CR, PR, or SD (reduction) after being treated with 2 cycles of anlotinib and trametinib.
5. No active brain metastases;
6. Age ≥18 years and ≤75 years;
7. ECOG PS score: 0 to 2;
8. Palliative radiotherapy must be completed 7 days before the first dose of study drug is administered;
9. The main organs function is normal, that is, the following criteria met:
10. Good hematopoietic function, defined as absolute neutrophil count ≥1.5×10^9 /L, platelet count≥100 ×10^9 /L, hemoglobin ≥90g/L [no blood transfusion or no erythropoietin (EPO) dependence within 7 days before enrollment]
11. Biochemical test results should meet the following criteria: BIL < 1.25 times the upper limit of normal value (ULN); ALT and AST < 2.5 × ULN; in case of liver metastases, ALT and AST < 5 × ULN; Cr ≤1.5×ULN or creatinine clearance (CCr) ≥60ml/min; Coagulation function is good, INR and PT ≤1.5 times ULN; if the subject is receiving anticoagulant treatment, PT should be within the prescribed range of use of anticoagulant drugs;
12. Women of child-bearing age should agree to take contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study and within 6 months after the study; non-breast-feeding patients whose serum or urinary pregnancy test should be negative; male patients should agree to take contraceptive measures during the study and within 6 months after the study.
13. Patients are voluntarily enrolled into the study, sign the informed consent form and have good compliance.

Exclusion Criteria:

1. Small cell lung cancer (including mixed small cell and non-small cell lung cancer);
2. Patients who have received previous treatment ≥ 4th lines of standard therapies.;
3. There are obvious bleeding symptoms or active autoimmune disease;
4. Patients with other driver mutation.
5. Patients with many factors affecting oral medication, such as dysphagia, gastrointestinal resection, chronic diarrhea and intestinal obstruction;
6. Patients who are known to have active brain metastases, spinal cord compression, carcinomatous meningitis, or brain or leptomeningeal disease diagnosed by CT or MRI at the time of screening;
7. Patients with severe and / or uncontrolled diseases, such as:
8. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmias; uncontrolled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
9. Active or uncontrolled serious infection;
10. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
11. Not completely controlled eye inflammation or eye infection, or any condition that may lead to the above-mentioned ocular diseases
12. Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
13. Routine urine test result indicates that urine protein ≥++, and 24-hour urine protein quantitation is confirmed to be > 1.0 g;
14. Active tuberculosis, etc.;
15. Uncontrolled hypercalcemia (> 1.5 mmol/L calcium ion or calcium > 12 mg/dL or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued diphosphate therapy;
16. Long-term unhealed wounds or fractures;
17. Patients who have a history of psychotropic drug abuse and cannot abstain from it or have mental disorders;
18. Patients who are known to have severe allergies (≥ grade 3) to active ingredients and any excipients of study drugs;
19. Patients who have other malignant tumors (except radical cervical carcinoma in situ, non-melanoma skin cancer, etc.) at the same time; patients who are evaluated by the investigator to have concomitant diseases that seriously endanger the safety of the patients or affect the patients completing the study.
20. The subjects or their sexual partners cannot or refuse to take effective contraceptive measures during the clinical trial.
21. Pregnant or breast-feeding women.
22. Patients who are allergic to any medicine or any ingredient; the patients with a history of treatments involving MEK inhibitors (trametinib, selumetinib, etc.) and RTKs inhibitors (anlotinib, sorafenib, apatinib, cabozantinib, etc.) were considered ineligible.
23. Patients in other situations who are evaluated by the investigator to be ineligible to be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
RP2D | up to 12 months
  recommended phase 2 dose
PFS | up to 18 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | up to 12 months
  objective response rate
OS | up to 24 months
  overall survival
DOR | up to 18 months
  duration of response
AEs | up to 24 months
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No